CLINICAL TRIAL: NCT03352219
Title: Reality Check: Evaluation of an HIV Risk Reduction Serial Drama for Black Youth
Brief Title: Reality Check: An HIV Risk Reduction Serial Drama
Acronym: RC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 822007; R34MH094207 (NIH)
Record Dates: First submitted 2017-11-17; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: HIV (Human Immunodeficiency Virus); Sexually Transmitted Diseases
Keywords: Human immunodeficiency virus; Sexually transmitted disease; African Americans; Young adults; Behavioral intervention; Entertainment-Education; Serial drama; Sexual behavior; HIV testing; Homophobia; Social cognitive theory
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Sexual Behavior; Homophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reality Check (Experimental): Received streamed 13-episode HIV risk reduction serial drama, Reality Check, developed based on Social Cognitive Theory integrated with findings from focus groups and community advisory boards. Each character has a behavioral trajectory related to HIV. For example, one character modeled negotiating condom use with his partner when she was against it. Messages in the serial drama showed that the characters had normative support for HIV testing and condom use. One character modeled a mastery experience when she overcame her fear and got tested for HIV. Homophobia is addressed when a mother discovers that her son is gay. Over the course of the episodes, the interweaving storylines play out, with all the characters eventually achieving their positive goals.
  Interventions: Behavioral: Reality Check
- Physical Activity Attention Control (Placebo Comparator): Received streamed physical activity promotion videos designed to control for Hawthorne effects, including special attention, consisting of a series of 13 videos from YouTube on physical activity and exercise. The videos, selected to be appropriate for African Americans 18 to 24 years of age, were tailored to be gender specific and hence varied between men and women. The videos focused on the importance of physical activity, coping strategies for lack of motivation to engage in physical activity, and other challenges faced in becoming more physically active, provided specific knowledge and skills regarding how to engage in aerobic and muscle-strengthening exercises, and model aerobic and muscle-strengthening exercises in a variety of settings.
  Interventions: Behavioral: Physical Activity Attention Control

INTERVENTIONS:
Behavioral: Reality Check
  Arms: Reality Check
Behavioral: Physical Activity Attention Control
  Arms: Physical Activity Attention Control

SUMMARY:
African Americans have considerably higher rates of HIV infections than do White, Hispanic, Asian, and Native Americans. African Americans accounted for 59% of all diagnoses of HIV infection among youth (13-24 years of age) in the United States. Young African Americans also have disproportionately high rates of other sexually transmitted infections (STIs). Therefore, the broad, long-term objective of this research is to identify interventions to reduce the risk of HIV and other STIs among young African Americans. Entertainment-education refers to narrative interventions designed to change behavior while providing entertainment. Several studies have evaluated the impact of media content on HIV risk behavior. One study found that exposure to an entertainment-education based HIV testing campaign was associated with increases in HIV testing among sexually active teens 12 months post exposure. Similarly, a radio soap opera called "Twende na Wakati" became the most popular television show in Tanzania and was highly successful in reducing the number of sexual partners and increasing condom use. A narrative video intervention study in STI clinic waiting rooms in three U.S. cities found a significant reduction in STI re-infection among patients visiting during months when the video was shown compared with patients visiting during months when it was not shown. Although these studies show that entertainment-education can be a promising medium for behavior change, none of them evaluated the efficacy of a tailored online entertainment-education intervention specifically designed for African American youth. To address this gap in the literature, this study tested the preliminary efficacy of an innovative, theory-based HIV risk-reduction serial drama intervention, Reality Check, specifically tailored to young African Americans. We used a randomized controlled trial, allocating African Americans 18 to 24 years of age to Reality Check, or an attention-control intervention promoting physical activity. Each intervention was delivered as a series of videos streamed online and accessible via any Internet-capable device. Participants completed surveys online at baseline, immediately post intervention, and 3 months post intervention. We hypothesized that, Reality Check would reduce condomless sex during the 3-month post-intervention period compared with the attention-matched control group, adjusting for baseline of the criterion.

DETAILED DESCRIPTION:
African Americans have considerably higher rates of HIV infections than do White, Hispanic, Asian, and Native Americans. African Americans accounted for 59% of all diagnoses of HIV infection among youth (13-24 years of age) in the United States. Young African Americans also have disproportionately high rates of other sexually transmitted infections (STIs). Therefore, the broad, long-term objective of this research is to identify interventions to reduce the risk of HIV and other STIs among young African Americans. Entertainment-education refers to narrative interventions designed to change behavior while providing entertainment. Several studies have evaluated the impact of media content on HIV risk behavior. One study found that exposure to an entertainment-education based HIV testing campaign was associated with increases in HIV testing among sexually active teens 12 months post exposure. Sabido and colleagues used "telenovelas" in Mexico to increase participation in a national literacy campaign and promote birth control use. Similarly, a radio soap opera called "Twende na Wakati" became the most popular television show in Tanzania and was highly successful in reducing the number of sexual partners and increasing condom use. A narrative video intervention study in STI clinic waiting rooms in three U.S. cities found a significant reduction in STI re-infection among patients visiting during months when the video was shown compared with patients visiting during months when it was not shown. Although these studies show that entertainment-education can be a promising medium for behavior change, none of them evaluated the efficacy of a tailored online entertainment-education intervention specifically designed for African American youth. To address this gap in the literature, this study tested the preliminary efficacy of an innovative, theory-based HIV risk-reduction serial drama intervention, Reality Check, specifically tailored to young African Americans and aimed at decreasing the frequency of condomless sex and promoting HIV testing among young adult African Americans. We used a randomized controlled trial, allocating African Americans 18 to 24 years of age to Reality Check, or an attention-control intervention promoting physical activity. Each intervention was delivered as a series of videos streamed online and accessible via any Internet-capable device (e.g., smartphone, laptop or tablet). This mode of delivery was well suited to young African Americans because high percentages of young African Americans own and use Internet enabled mobile phones as their primary way to consume online content. We recruited participants through Facebook and Instagram, flyers posted on college campuses, college mailing lists, and referrals from participants. Participants completed surveys online at baseline, immediately post intervention, and 3 months post intervention. We hypothesized that, Reality Check would reduce the frequency of condomless sex during the 3-month post-intervention period compared with the attention-matched control group, adjusting for baseline of the criterion.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as black or African American, had a Facebook ID, had a smartphone with access to the Internet, and reported having sexual intercourse in the previous 90 days

Exclusion Criteria:

* None

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Frequency of condomless sexual intercourse | 3 months post-intervention
  The number of times the participant had sex without using a condom in the past 90 days

SECONDARY OUTCOMES:
Frequency of condom use | 3 months post-intervention
  Rated frequency of condom use in the past 90 days
Consistent (100%) condom use | 3 months post-intervention
  A binary variable indicating whether the participants used a condom 100% of the time during sex in the past 90 days
Frequency of sexual intercourse | 3 months post-intervention
  The number of times the participant had sexual intercourse in the past 90 days
HIV testing | 3 months post-intervention
  A binary variable indicating whether the participant reported being tested for HIV in the past 3 months
Homophobia | Immediately post-intervention
  Negative attitude toward homosexuals
Homophobia | 3 months post-intervention
  Negative attitude toward homosexuals
AIDS-related stigma | Immediately post-intervention
  Negative attitudes toward AIDS
AIDS-related stigma | 3 months post-intervention
  Negative attitudes toward AIDS

CONTACTS AND LOCATIONS:
Overall Officials: John B Jemmott III, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Annenberg School for Communication, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No